CLINICAL TRIAL: NCT00787358
Title: A Randomized, Double-Blind, Placebo Controlled Proof-of-Concept Study Investigating the Safety and Efficacy of ZT-031 on Hip Fracture Healing in Men and Postmenopausal Women With Intertrochanteric Fracture of the Hip
Brief Title: A Proof-of-Concept Study Investigating the Safety and Efficacy of ZT-031 on Hip Fracture Healing in Men and Postmenopausal Women
Acronym: SHIFT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in company direction
Sponsor: Zelos Therapeutics (Industry)
Responsible Party: Dr. David S. Krause, Chief Medical Officer, Zelos Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OC-018
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Hip Fracture
Keywords: osteoporosis; intertrochanteric; hip fracture; compression hip screw; surgical fixation
MeSH Terms: conditions — Hip Fractures; Osteoporosis | interventions — ZT-031

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZT-031 (Active Comparator)
  Interventions: Drug: ZT-031
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ZT-031 — 80 ul subcutaneous injection per day
  Arms: ZT-031
Other: placebo — 80 ul daily subcutaneous injection of vehicle only
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test if an experimental drug called ZT-031 can help men over 30 years or post-menopausal women over 55 years of age with certain types of hip fracture to heal better or faster following surgery and to determine if ZT-031 is safe for patients with fractures. To be allowed in the study you have to have a type of hip fracture that requires surgery that is being studied (intertrochanteric fracture). You must also otherwise be in good health, with no serious diseases such as cancer, neurologic disease, other bone disease, liver, heart or kidney disease. You must be able to inject yourself every day with the study medication using an injection pen, like that used for insulin injections.

ELIGIBILITY:
Inclusion Criteria

Subjects are required to meet all of the following criteria for inclusion in the study:

1. Signed Institutional Review Board (IRB)/Research Ethics Board (REB)-approved informed consent form (ICF).
2. Sustained an unstable low energy intertrochanteric (Evans Type II or higher) hip fracture within 7 days prior to planned surgery date. Low energy is defined as a fracture that occurs spontaneously or from a fall from a stationary height of ≤ 1 meter (3 feet) or missing one to three steps.
3. Women ≥ 55 years of age and men ≥ 30 years of age of any race. If female, subjects must be post-menopausal for at least 5 years and weigh ≥ 110 lbs or 50 kg.
4. Subjects who are expected to undergo or have recently undergone (within two weeks) open or closed repair of the fracture requiring a CHS.
5. By history, the subject was at least household ambulatory prior to hip fracture.
6. Serum calcium level within the normal range when corrected for albumin. Corrected calcium (mg/dL) = Serum Ca (mg/dL) + 0.8 x (4.0 - albumin [g/dL])
7. Able and willing to comply with all protocol procedures.
8. Cognitive, visual, auditory and physical abilities adequate to undertake assessments.
9. Availability of a care partner to administer injections or demonstrated ability to self-administer injections. Subjects planning to self-administer study drug will need to show that they will be capable of accurately self-injecting study drug in rotating quadrants of the abdomen, in the opinion of the Investigator.
10. Clinically acceptable medical history and physical examination, according to the judgment of the Investigator.
11. Laboratory results within normal ranges or, if abnormal, considered by the Investigator as not clinically significant for the well-being of the subject or for the purpose of the study.

    The following additional criteria are required for randomization and dosing with ZT-031 or placebo to occur:
12. The most recent value for 25-hydroxy Vitamin D (25OHD) must be at or above the lower limit of normal (LLN) for the laboratory reference range of the testing method used for determination of 25OHD. NOTE: Randomization should be delayed until it is known that 25OHD is ≥ LLN.
13. The most recent value for intact PTH must be ≤ ULN for the laboratory reference range.
14. Randomization and dosing must occur within 2 weeks post-op. Exclusion Criteria

Subjects who meet any of the following conditions are excluded from this clinical study:

1. Previous fracture(s) or bone or joint surgery in the currently fractured site
2. Intertrochanteric fracture with reverse obliquity
3. Pathologic fracture: A fracture occurring at a site of metabolic bone disease (other than osteoporosis) or a benign or malignant tumor
4. Presence of a concurrent disease known to affect bone metabolism other than post-menopausal osteoporosis, including but not limited to hyperparathyroidism, hyperthyroidism, osteogenesis imperfecta, abnormalities of serum calcium, Paget's disease, or osteomalacia
5. History of rheumatoid arthritis
6. Any significant neurologic disease including but not limited to any dementing illness or other neurodegenerative disease, cerebrovascular disease, epilepsy or undiagnosed syncope
7. Unstable or clinically significant cardiovascular disease resulting in:

   1. Hemodynamic instability manifested as hypotension unresponsive to intravenous fluids
   2. Uncontrolled hypertension requiring administration of parenteral therapy.
8. Renal disease, defined by:

   1. Creatinine level of >2.0 mg/dL
   2. Urolithiasis or nephrolithiasis in the last 2 years
9. Hepatic disease or insufficiency, defined by liver function tests (ALT, AST or GGT) > 3 times the ULN or bilirubin > 34 mmol/L or 2.0 mg/dL
10. Currently receiving treatment for cancer
11. History of external beam radiation to the skeleton or a radiation therapy implant device
12. Presence of substance abuse, including alcohol, within 1 year of Screening
13. Current or previous use of any PTH compound, including ZT-031
14. Use of any investigational compound within 4 weeks of Screening, or within 5 half-lives of compound, whichever is longer
15. Use of any bone substitutes, osteobiologics or any fracture healing drug.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Compression hip screw (CHS) migration: the difference in the tip apex distance (TAD) post-operatively to that at Visit 7/Week 16 | 16 weeks

SECONDARY OUTCOMES:
Screw barrel impaction distance | 16 weeks
Screw cut-out and/or other hardware failure | 16 weeks
Incidence of fracture non-union | 16 weeks
Need for surgical revision with or without hardware removal | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- J. Edward Puzas, Rochester, New York, United States